CLINICAL TRIAL: NCT07150845
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study Evaluating the Efficacy and Safety of EVO756 in Adults With Atopic Dermatitis
Brief Title: Phase 2b Study of EVO756 in Adults With Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Evommune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVO756-AD001
Record Dates: First submitted 2025-08-28; First posted 2025-09-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Atoptic Dermatitis
Keywords: atopic dermatitis; eczema; itch
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose 1 (Experimental): Orally administered EVO756, Dose 1
  Interventions: Drug: EVO756
- Dose 2 (Experimental): Orally administered EVO756, Dose 2
  Interventions: Drug: EVO756
- Dose 3 (Experimental): Orally administered EVO756, Dose 3
  Interventions: Drug: EVO756
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: EVO756 — Dose 1
  Arms: Dose 1
Drug: EVO756 — Dose 2
  Arms: Dose 2
Drug: EVO756 — Dose 3
  Arms: Dose 3
Drug: Placebo control — Placebo control
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of different doses of EVO756 in adults with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic AD that has been present for ≥6 months
* Validated-Investigator's Global Assessment score of ≥3
* EASI of ≥16
* BSA of AD involvement of ≥10%

Exclusion Criteria:

* Any clinically significant abnormality in laboratory evaluations, physical examinations, vital signs, or ECG at Screening
* Use of certain medications
* Presence of skin comorbidities or other condition(s) that may interfere with study assessments
* Significant AD flare, in the opinion of the Investigator, within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage change in Eczema Area and Severity Index (EASI) from Baseline | Week 12

SECONDARY OUTCOMES:
Percentage change in EASI from Baseline | Weeks 2, 4, and 8
Mean changes in EASI from Baseline | Week 2, 4, 8, and 12
Proportion of subjects with EASI-50, EASI-75, and EASI-90 from Baseline | Weeks 2, 4, 8, and 12
Mean and absolute changes in validated Investigator Global Assessment (vIGA) score from Baseline | Weeks 2, 4, 8, and 12
Proportion of subjects achieving a vIGA score of 0,1 with at least a 2-point reduction from Baseline | Weeks 2, 4, 8, and 12
Mean and percentage change from Baseline in the pruritus-NRS score | Weeks 2, 4, 8, and 12
Proportion of subjects achieving a 4-pt reduction in the pruritus-NRS score from Baseline | Week 2, 4, 8, and 12
Mean and percentage changes from Baseline in Body Surface Area (BSA) of affected area | Weeks 2, 4, 8, and 12
Occurrence of treatment emergent adverse events (TEAE) and serious adverse events (SAE) | through Week 14

CONTACTS AND LOCATIONS:
Locations (24):
- United States (20):
  - Center for Dermatology Clinical Research, Fremont, California
  - Metropolis Dermatology - Downtown Los Angeles, Los Angeles, California
  - Skin and Beauty Center, Pasadena, California
  - Skin Care Research, LLC, Boca Raton, Florida
  - Driven Research, LLC, Coral Gables, Florida
  - Skin Care Research - Hollywood Dermatology, Hollywood, Florida
  - TrueBlue Clinical Research, Tampa, Florida
  - DS Research, Clarksville, Indiana
  - Equity Medical, Bowling Green, Kentucky
  - Aesthetic and Dermatology Center, Rockville, Maryland
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Empire Dermatology, East Syracuse, New York
  - Equity Medical, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - International Clinical Research - Murfreesboro, Murfreesboro, Tennessee
  - Stryde Research, Lewisville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
- New Zealand (4):
  - Pacific Clinical Research Network (PCRN) - Christchurch, Christchurch Central City, Christchurch
  - Optimal Clinical Trials, Auckland, NZL
  - Clinical Trials NZ Limited, Hamilton, NZL
  - Momentum Clinical Research Lower Hutt, Lower Hutt, NZL